CLINICAL TRIAL: NCT00148291
Title: Phase III Study of Docetaxel Vs Vinorelbine in Elderly Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West Japan Thoracic Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJTOG9904
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2006-01-06 (Estimated); Status verified 2005-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Vinorelbine

INTERVENTIONS:
Drug: Patients were randomized to receive either docetaxel 60 mg/m2 on day 1 or vinorelbine 25 mg/m2 on days 1and 8, repeated every 21 days over four cycles.

SUMMARY:
Vinorelbine is currently the standard treatment for elderly patients with advanced non-small cell lung cancer (NSCLC). Docetaxel has also shown promising results against elderly patients in phase II studies. We conducted a randomized phase III trial to evaluate whether docetaxel provided better overall survival than vinorelbine in elderly patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

Chemotherapy- and radiotherapy-naïve patients with histologically or cytologically diagnosis of stage IIIB or IV NSCLC and who were ≧ 70 years old with measurable or assessable disease were eligible for this trial. They had to have a life expectancy of at least 3 months. Additional entry criteria were as follows: (a) a performance status (PS) 0 to 2 on the Eastern Cooperative Oncology Group scale; (b) adequate function of bone marrow (leukocyte count ≧ 4,000/μL, absolute neutrophil count ≧ 2,000/μL, hemoglobin concentration ≧ 9.5 g/dL, platelet count ≧ 100,000/μL), kidney (serum creatinine ≦ 1.2 mg/dL), liver (total bilirubin ≦ 1.5 times the institutional upper limits of normal, transaminase of AST and ALT ≦ 2.5 times the institutional upper limits of normal).

Exclusion Criteria:

Patients with symptomatic brain metastasis or apparent dementia were ineligible. Patients with active concomitant malignancy, massive pleural effusion or ascites, active infection, severe heart disease, grade 2 or higher ECG abnormality, uncontrolled diabetes mellitus, ileus, pulmonary fibrosis, diarrhea, and a bleeding tendency were excluded.-

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Overall Officials: Shinzoh Kudoh, MD, Principal Investigator — West Japan Thoracic Oncology Group

REFERENCES:
- See also: Related Info — http://www.wjtog.org/